CLINICAL TRIAL: NCT00974571
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Investigating the Clinical Effects of Montelukast in Patients With Perennial Allergic Rhinitis
Brief Title: Montelukast in Perennial Allergic Rhinitis - 2001-2002 Study (0476-246)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-246; MK0476-246; 2009_659
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast sodium
- 2 (Active Comparator): cetirizine
  Interventions: Drug: Comparator: cetirizine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: montelukast sodium — montelukast 10 mg tablet orally once daily at bedtime for 6 weeks
  Arms: 1
Drug: Comparator: cetirizine — cetirizine 10 mg tablet orally once daily at bedtime for 6 weeks
  Arms: 2
Drug: Comparator: placebo — placebo tablet orally once daily at bedtime for 6 weeks
  Arms: 3

SUMMARY:
This study will assess the ability of montelukast to improve the signs and symptoms of perennial allergic rhinitis compared to placebo. Cetirizine is included in the study as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented clinical history of perennial allergic rhinitis
* Patient is a nonsmoker
* Patient is in good general health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is <8 weeks postpartum or is breast-feeding
* Patient is a current or past abuser of alcohol or illicit drugs

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1365 (Actual)
Dates: Start 2001-11; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Philip G, Williams-Herman D, Patel P, Weinstein SF, Alon A, Gilles L, Tozzi CA, Dass SB, Reiss TF. Efficacy of montelukast for treating perennial allergic rhinitis. Allergy Asthma Proc. 2007 May-Jun;28(3):296-304. doi: 10.2500/aap.2007.28.3000. PMID 17619558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 study sites in the United States
  Primary Therapy: Nov-2001 to May-2002
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime rhinitis symptoms score during the run-in period were excluded from randomization.
Groups:
- Montelukast 10 mg: Montelukast 10-mg film-coated tablet and cetirizine matching-image placebo tablet orally once daily at bedtime for 6 weeks.
- Cetirizine 10 mg: Montelukast matching-image placebo tablet and cetirizine 10-mg tablet orally once daily at bedtime for 6 weeks.
- Placebo: Montelukast matching-image placebo tablet and cetirizine matching-image placebo tablet orally once daily at bedtime for 6 weeks.
Period: Overall Study
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Started | 630 | 122 | 613
Completed | 562 | 106 | 530
Not Completed | 68 | 16 | 83
Not completed — Adverse Event | 31 | 4 | 27
Not completed — Lack of Efficacy | 3 | 2 | 9
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Protocol Violation | 13 | 4 | 18
Not completed — Withdrawal by Subject | 14 | 5 | 16
Not completed — Patient Moved | 1 | 0 | 1
Not completed — Other | 4 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo | Total
Number analyzed (Participants) | 630 | 122 | 613 | 1365
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (12.87) | 36.3 (13.67) | 35.3 (13.17) | 35.4 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 419 | 85 | 418 | 922
  Male | 211 | 37 | 195 | 443
Composite Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Composite Symptoms Scores were computed as the average of the Daytime Nasal Symptoms Scores [Score 0 (best) to 3 (worst)] and Nighttime Symptoms Scores [Score 0 (best) to 3 (worst)].
  Scores on a scale | 1.86 (0.44) | 1.89 (0.43) | 1.82 (0.45) | 1.85 (0.44)
Daytime Nasal Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Patients were asked to rate each of 4 nasal symptoms of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual nasal symptom scores was reported as the Daytime Nasal Symptoms Score.
  Scores on a scale | 2.08 (0.40) | 2.13 (0.37) | 2.07 (0.40) | 2.08 (0.40)
Nighttime Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Patients were asked to rate each of 3 symptoms of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings daily on a 4-point scale [Score 0 (best) to 3 (worst)], and the average score of the 3 symptoms was reported as the Nighttime Symptoms Score.
  Scores on a scale | 1.63 (0.62) | 1.65 (0.61) | 1.58 (0.62) | 1.61 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score
Description: Mean change from baseline in Daytime Nasal Symptoms score.
  Patients were asked to rate each nasal symptom of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
Time Frame: Baseline and first 4 weeks of a 6-week treatment period
Population: All patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Number analyzed (Participants) | 626 | 120 | 609
Scores on a scale | -0.39 [-0.43 to -0.36] | -0.45 [-0.54 to -0.37] | -0.36 [-0.39 to -0.32]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score
Description: Mean change from baseline in Nighttime Symptoms Score.
  Patients were asked to rate each symptom daily on a 4-point scale [Score 0 (best) to 3 (worst)], and the average score of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings was reported as the Nighttime Symptoms Score.
Time Frame: Baseline and first 4 weeks in 6-week treatment period
Population: All patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Number analyzed (Participants) | 626 | 120 | 609
Scores on a scale | -0.28 [-0.32 to -0.25] | -0.30 [-0.38 to -0.23] | -0.26 [-0.29 to -0.22]

3. Secondary Outcome: Mean Change From Baseline in Composite Symptoms Score
Description: Composite Symptoms Scores were computed as the average of the Daytime Nasal Symptoms Scores [Score 0 (best) to 3 (worst)]. and Nighttime Symptoms Scores collected [Score 0 (best) to 3 (worst)].
Time Frame: Baseline and first 4 weeks in 6-week treatment period
Population: All patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score 0 (best) to 3 (worst)
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Number analyzed (Participants) | 626 | 120 | 609
Score 0 (best) to 3 (worst) | -0.34 [-0.37 to -0.31] | -0.38 [-0.45 to -0.31] | -0.30 [-0.34 to -0.27]

4. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the patient, administered at week 4 of the study (or upon discontinuation) using a 7-point scale [Score 0 (best) to 6 (worst)], of the change in symptoms as compared to the beginning of the study.
Time Frame: End of the first 4 weeks in 6-week treatment period
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle. Since only 1 measurement was obtained during the treatment period, no missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Number analyzed (Participants) | 617 | 117 | 602
Scores on a scale | 2.22 [2.11 to 2.32] | 2.15 [1.92 to 2.38] | 2.41 [2.30 to 2.51]

5. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the physician, administered at week 4 of the study (or upon discontinuation) using a 7-point scale [Score 0 (best) to 6 (worst)], of the change in symptoms as compared to the beginning of the study.
Time Frame: End of the first 4 weeks in 6-week treatment period
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Number analyzed (Participants) | 603 | 115 | 583
Scores on a scale | 2.26 [2.16 to 2.36] | 2.20 [1.99 to 2.42] | 2.33 [2.23 to 2.43]

ADVERSE EVENTS:
Time Frame: During the 6 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy
Description: The number of patients listed in the Adverse Event tables (613 in the placebo group, 630 in the montelukast group, and 122 in the cetirizine group) is the number of patients who received study treatment.
Arm/Group | Montelukast 10 mg | Cetirizine 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/630 | 0/122 | 3/613
Other Adverse Events (participants affected / at risk) | 85/630 | 16/122 | 65/613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 10 mg (N=630) | Cetirizine 10 mg (N=122) | Placebo (N=613)
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Unstable Angina (Cardiac disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 10 mg (N=630) | Cetirizine 10 mg (N=122) | Placebo (N=613)
Upper Respiratory Infection (Infections and infestations) | 41 | 8 | 34
Headache (Nervous system disorders) | 47 | 8 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.